CLINICAL TRIAL: NCT05791318
Title: A Phase 1, Randomized, Triple-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of the Monoclonal Antibody VYD222 in Healthy Adult Participants
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of the Monoclonal Antibody VYD222 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invivyd, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: VYD222-1-001
Record Dates: First submitted 2023-03-16; First posted 2023-03-30 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, triple blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 10 total participants Cohort 1. 8 participants on VYD222 2 participants on placebo
  Interventions: Drug: VYD222; Other: Placebo
- Cohort 2 (Experimental): 10 total participants Cohort 2. 8 participants on VYD222 2 participants on placebo
  Interventions: Drug: VYD222; Other: Placebo
- Cohort 3 (Experimental): 10 total participants Cohort 3. 8 participants on VYD222 2 participants on placebo
  Interventions: Drug: VYD222; Other: Placebo

INTERVENTIONS:
Drug: VYD222 — Monoclonal antibody
Other: Placebo — Matching Placebo
  Other Names: 0.9% sodium chloride

SUMMARY:
A study to investigate the safety, tolerability, and pharmacokinetics of the monoclonal antibody VYD222 in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, randomized, triple blind, single escalating dose study to evaluate the safety and tolerability of VYD222, a monoclonal antibody targeting SARS-CoV-2, in healthy adult volunteers.

The primary objective is to evaluate the safety and tolerability of multiple dose levels of VYD222 after a single administration in healthy participants. The secondary objective is to evaluate the plasma pharmacokinetics and immunogenicity of VYD222 after administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index 18.5 to 32.0 kg/m2, inclusive.
* Negative for current SARS-CoV-2 infection by rapid antigen test on Day -1.
* Is seropositive to N and/or S SARS-CoV-2 antigens at Screening.
* For participants assigned female sex at birth: Is not of childbearing potential OR is of childbearing potential and practicing highly effective contraception.
* Is able and willing to provide written informed consent.
* NOTE: Other protocol defined inclusion/exclusion criteria apply

Exclusion Criteria:

* Intends to receive a COVID-19 vaccine/booster within 3 months of Day 1.
* Is pregnant, breastfeeding, or seeking pregnancy while on study.
* Has a history of a malignancy (or active malignancy), except for participants with basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix who have been treated and cured.
* Has had any symptoms of acute respiratory illness (e.g., cough, shortness of breath, sore throat, fatigue, loss of smell, fever), or other febrile illness within 2 weeks prior to dosing.
* Has evidence of active infection with HIV, HBV, or HCV.
* Has donated more than 500 mL of blood within 60 days before the scheduled dose of study drug.
* Had major surgery within 30 days prior to study drug dosing or planned surgeries within 12 months after planned study drug dosing.
* Received any investigational drug or biologic within 30 days or 5 half-lives (whichever is longer) prior to Screening or planned administration of any investigational drug or biologic during the study period.
* Received immunoglobulin or blood products within 6 months prior to Screening.
* Previously received a mAb within 6 months or 5 half-lives (whichever is longer) prior to Screening.
* NOTE: Other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAEs (including AEs and SAEs) | Through 12 Months

SECONDARY OUTCOMES:
Incidence of ADAs against VYD222 | 12 Months
Assessment of PK Parameter: area under the concentration-time curve from time zero extrapolated to infinity for VYD222 | 12 Months
Assessment of PK Parameter: area under the concentration-time curve from time zero to the last measurable concentration for VYD222 | 12 Months
Assessment of PK Parameter: area under the concentration-time curve from time zero to t for VYD222 | 12 Months
Assessment of PK Parameter: Cmax (maximum serum concentration) | 12 Months
Assessment of PK Parameter: Tmax (time to reach maximum serum concentration) | 12 Months
Assessment of PK Parameter: Clearance of VYD222 | 12 Months
Assessment of PK Parameter: Half-life of VYD222 | 12 Months
Assessment of PK Parameter: volume of distribution at steady state of VYD222 | 12 Months
Assessment of PK Parameter: volume of distribution during terminal phase of VYD222 | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Joondalup, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No